CLINICAL TRIAL: NCT06161285
Title: Association of Dysbiosis and Immune Response in Bronchiolitis in Under 12 Months -Old Infants
Acronym: BRONCHOBIOTE
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Infectious Diseases Models for Innovative Therapies center (Unknown)
Responsible Party: Sponsor
Other Study IDs: APHP231177; 2023-A01688-37 (Other: IDRCB)
Record Dates: First submitted 2023-11-30; First posted 2023-12-07 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-01

CONDITIONS: Bronchiolitis
Keywords: Newborns; Dysbiosis; respiratory syncytial virus (RSV)
MeSH Terms: conditions — Bronchiolitis; Dysbiosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Severe bronchiolitis: venous blood samples. Buccal, nasopharyngeal and rectal swabs
  Interventions: Other: Sampling
- Non-hospitalized bronchiolitis: Capillary blood samples. Buccal, nasopharyngeal and rectal swabs
  Interventions: Other: Sampling
- Bronchiolitis ihospitalized in ICU: Capillary blood samples. Buccal, nasopharyngeal and rectal swabs

INTERVENTIONS:
Other: Sampling — Single-time sampling of respiratory virus-infected children
  Groups: Non-hospitalized bronchiolitis; Severe bronchiolitis

SUMMARY:
Acute bronchiolitis is a common disease in children under the age of two, caused mainly by the respiratory syncytial virus (RSV). Furthermore, given the same medical history, it is still very difficult to predict the course and severity of the infection at the onset of symptoms, Some studies have highlighted the importance of the microbiota (intestinal, oral or nasopharyngeal) and of the immune response to RSV in children, We will include 80 children under 2 years old with hospitalized bronchiolitis and non-hospitalized bronchiolitis. Oral, nasal and stool samples will be taken to study the various microbiota in search of dysbiosis. A capillary blood sample will be taken for immune studies.

ELIGIBILITY:
Inclusion Criteria:

* Infants <12 months
* With bronchiolitis during RSV epidemic season
* No chronic illness
* No bronchiolitis medical history
* Signed consent from parents or legal guardians

Exclusion Criteria:

* Chronic respiratory illness
* Medical history of bronchiolitis or newborn asthma
* Treatment with immunosuppressants
* Patient with no social security affiliation

Ages: 1 Day to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Bronchiolitis in patient under 12 months old
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-12-06 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Dysbiosis | Inclusion
  comparison of the quantitative and qualitative composition of bacteria (alpha diversity, beta diversity, Shannon and Simpson index) in the digestive and nasopharyngeal microbiota

SECONDARY OUTCOMES:
Measurement of innate and adaptive responses by quantification of cytokines and chemokines in plasma | inclusion
  Inflammatory/regulatory cytokines (IL1->17, IL-10, TGF-b, EGF, FGF-2, IFN-alpha, IFN-gamma, IFN-beta, MCRP-1 MCP-3, TNF-alpha...), cytokines of adaptative response (Th1, Th17, Th2 and/or Treg), markers of inflammatory response (interferon, TNFa, …), quantified by Luminex
Identifying the mRNA profile in blood samples and nasal swabs | inclusion
  mRNA will be identified by using RNA-Seq (Illumina)
Sequencing viral strains for mutation | Inclusion
  Typing of respiratory syncytial virus-A (RSV-A) and B (RSV-B) and sequencing of strains (Amplicons)
Comparison of respiratory syncytial virus (RSV) antibodies levels on newborn screening specimen and on capillary swab during infection | Birth, Inclusion
  Levels of RSV antibodies will be measured and compared between newborn screening specimen and capillary swab during infection
Study the load of Streptococcus pneumoniae (Sp) in RSV infections. | Inclusion
  Compare the serotypic profiles of pneumococcus (Sp) present during RSV infections

CONTACTS AND LOCATIONS:
Overall Officials: Etienne BIZOT, Doctor, Principal Investigator — AP-HP Hôpital Antoine Beclere
Locations (3):
- France (3):
  - APHP, Antoine Béclère Hospital, Clamart
  - AP-HP,Raymond Poincaré Hospital, Garches
  - Réanimation médico-chirurgicale Necker, Paris

IPD SHARING:
Plan to Share IPD: No